CLINICAL TRIAL: NCT02820649
Title: Protective Effects of Exercise Training on Endothelial Dysfunction Induced by Total Sleep Deprivation in Healthy Subjects
Brief Title: Protective Effects of Exercise Training
Acronym: SOMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Collaborators: Cetre du sommeil et de la vigilance, APHP (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PDH-1-SMO-2-508; 2014_A01103-44 (Other: IDRCB ANSM)
Record Dates: First submitted 2016-06-23; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Sleep Deprivation
Keywords: Exercise training; Endothelial function
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (Experimental): 7 weeks of exercise training
  Interventions: Other: Sleep deprivation
- Control (Sham Comparator): Sedentary group
  Interventions: Other: Sleep deprivation

INTERVENTIONS:
Other: Sleep deprivation — 40 hours of continuous wakefullness

SUMMARY:
Rationale. Sleep loss is a risk factor for cardiovascular events mediated through endothelial dysfunction.

Objective. To determine if 7 weeks of exercise training can limit cardiovascular dysfunction induced by total sleep deprivation (TSD) in healthy young men.

Methods: 16 subjects will be examined during 40-h TSD, both before and after 7 weeks of interval exercise training. Vasodilatation induced by ACh, insulin and heat (42°C) as well as pulse wave velocity (PWV), blood pressure and heart rate (HR) will be assessed at baseline, during TSD, and after one night of sleep recovery. Biomarkers of endothelial activation, inflammation, and hormones will bemeasured from morning blood samples at 07:00

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Men
* 18 - 35 yrs

Exclusion Criteria:

* Consumming 400 mg of caffeine per day,
* Body mass index (BMI) greater than 30 kg/m²,
* Taking medication.
* Excessive daytime somnolence (Epworth Sleepiness Scale >9)
* Sleep complaints (Pittsburgh Sleep Quality Index >5)
* Inability to be considered as an intermediate chronotype on the Horne and Ostberg questionnaire (score <31 or >69)
* Traines subject (Ricci Gagnon questionnaire >35)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
ACh induced Vasodilation during TSD | Up to 09:00 during sleep deprivation (i.e. after 26 hours of wakefulness)
  Cutaneous vasodilation (in % Baseline) induced by local application of Acethylcholine

SECONDARY OUTCOMES:
Insuline Vasodilation | Up to 09:00 during the sleep deprivation day and the recovery day
  Cutaneous vasodilation (in % Baseline) induced by local application of insulin
Heat vasodilation | Up to 9:00 during the sleep deprivation day and during the recovery day
  Cutaneous vasodilation (in % Baseline) induced by local application of heat (42°C)
Inflammation | Up to 7:00 during the sleep deprivation day and during the recovery day.
  Plasma levels of inflammatory marquers (TNF-alpha, IL1beta...)
blood pressure | Every 3 hours during the 40 hours of wakefullness (i.e. total sleep deprivation)
  Mean, systolic and diastolic blood pressure
PWV | Up to 09:00 during the sleep deprivation day
  Pulse wave velovity evaluated by echography

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sauvet F, Drogou C, Bougard C, Arnal PJ, Dispersyn G, Bourrilhon C, Rabat A, Van Beers P, Gomez-Merino D, Faraut B, Leger D, Chennaoui M. Vascular response to 1 week of sleep restriction in healthy subjects. A metabolic response? Int J Cardiol. 2015;190:246-55. doi: 10.1016/j.ijcard.2015.04.119. Epub 2015 Apr 16. PMID 25932797
- [Background] Arnal PJ, Drogou C, Sauvet F, Regnauld J, Dispersyn G, Faraut B, Millet GY, Leger D, Gomez-Merino D, Chennaoui M. Effect of Sleep Extension on the Subsequent Testosterone, Cortisol and Prolactin Responses to Total Sleep Deprivation and Recovery. J Neuroendocrinol. 2016 Feb;28(2):12346. doi: 10.1111/jne.12346. PMID 26647769
- [Background] Arnal PJ, Sauvet F, Leger D, van Beers P, Bayon V, Bougard C, Rabat A, Millet GY, Chennaoui M. Benefits of Sleep Extension on Sustained Attention and Sleep Pressure Before and During Total Sleep Deprivation and Recovery. Sleep. 2015 Dec 1;38(12):1935-43. doi: 10.5665/sleep.5244. PMID 26194565
- [Derived] Sauvet F, Arnal PJ, Tardo-Dino PE, Drogou C, Van Beers P, Bougard C, Rabat A, Dispersyn G, Malgoyre A, Leger D, Gomez-Merino D, Chennaoui M. Protective effects of exercise training on endothelial dysfunction induced by total sleep deprivation in healthy subjects. Int J Cardiol. 2017 Apr 1;232:76-85. doi: 10.1016/j.ijcard.2017.01.049. Epub 2017 Jan 5. PMID 28089456